CLINICAL TRIAL: NCT05903820
Title: The Effect of Low-dose Rhythmic 17-β-estradiol Administration on Bone Turnover in Postmenopausal Women
Brief Title: Rhythmic Estradiol and Bone Health
Acronym: REBEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Peter H. Bisschop, Principal Investigator, Amsterdam UMC, location AMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL83336.018.23
Record Dates: First submitted 2023-05-15; First posted 2023-06-15 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-07

CONDITIONS: Osteoporosis Risk; Menopause
MeSH Terms: interventions — Ortho Evra; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Continuous estradiol 50 mcg/day (Active Comparator): The continuous standard-dose 17-β-estradiol group will receive the standard therapy for prevention of osteoporosis. A transdermal patch that releases 50ug/24 hrs of 17-β-estradiol will be administered continuously during the 16 weeks of treatment.
  Interventions: Drug: Estradiol patch; Drug: Progesterone
- Continuous estradiol 25 mcg/day (Active Comparator): The continuous low-dose 17-β-estradiol group will receive a transdermal patch that releases 25ug/24 hrs of 17-β-estradiol administered continuously during the 16 weeks of treatment.
  Interventions: Drug: Estradiol patch; Drug: Progesterone
- Rhythmic estradiol 25-50 mcg/day (Experimental): The rhythmic 17-β-estradiol group will receive a transdermal patch for two weeks that releases 25ug/24hrs of 17-β-estradiol, and a patch of 50ug/24hrs for 2 weeks in each 4-week cycle.
  Interventions: Drug: Estradiol patch; Drug: Progesterone

INTERVENTIONS:
Drug: Estradiol patch — Transdermal patch of estradiol
  Other Names: transdermal17-beta-estradiol
Drug: Progesterone — Oral progesterone capsules 100mg/day
  Other Names: micronized progesterone

SUMMARY:
The goal of this randomized-controlled trial is to compare the effect of rhythmic estrogen treatment to continuous estrogen treatment on bone turnover in healthy postmenopausal women. The main question it aims to answer are:

• Does rhythmic estrogen lead to increased bone formation in healthy postmenopausal women, compared to continuous estrogen?

Participants will receive one of the following treatments for a duration of 16 weeks:

- Rhythmic estradiol: Alternating 4-week cycles consisting of transdermal 17-β-estradiol 25μg/24hrs for two weeks, followed by two weeks of transdermal 17-β-estradiol 50μg/24hrs. Estradiol therapy will be combined with continuous oral micronized progesterone 100mg once daily.

* Low-dose continuous estradiol: Continuous transdermal 17-β-estradiol 25μg/24hrs, combined with continuous oral micronized progesterone 100mg daily once daily.
* Standard-dose continuous estradiol: Continuous transdermal 17-β-estradiol 50μg/24hrs, combined with continuous oral micronized progesterone 100mg daily once daily.

If there is a comparison group: Researchers will compare rhythmic estradiol to continuous estradiol to see if rhythmic estradiol improves bone formation in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, defined as final menstrual cycle more than 1 years prior to inclusion and FSH>30 IU/L
* Final menstrual cycle < 10 years prior to inclusion

Exclusion Criteria:

* Contra-indication for estrogen and/or progesterone therapy
* First-grade family member with inherited thrombophilia or history of venous thromboembolism under the age of 60 years
* Hysterectomy
* Premature menopause (menopause age <40 years)
* Known hypersensitivity to the excipients in the estradiol patch or progesterone capsule
* Hormonal contraception or hormone replacement therapy use (estradiol with or without progesterone) in the past 12 months
* Presence or history of any clinically relevant metabolic, endocrinological, hepatic, renal, cardiovascular, gastrointestinal, or respiratory conditions, history of bone disease or bone marrow disease, known vitamin D deficiency (25-OH vitamin D <30 nmol/L)
* Recent fracture (<12 months)
* BMI <20 or BMI ≥30
* Use of drugs including herbal medicine known to affect bone metabolism (e.g. corticosteroids) or to interfere with cytochrome P450 enzyme (CYP) pathways. Exceptions are occasional use of paracetamol, ibuprofen, acetylsalicylic acid or topical medication

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Serum P1NP | The difference in P1NP between treatment arms after 2 weeks
  The interaction between treatment and time on serum P1NP
Serum P1NP | The difference in P1NP between treatment arms after 4 weeks
  The interaction between treatment and time on serum P1NP
Serum P1NP | The difference in P1NP between treatment arms after 6 weeks
  The interaction between treatment and time on serum P1NP
Serum P1NP | The difference in P1NP between treatment arms after 8 weeks
  The interaction between treatment and time on serum P1NP
Serum P1NP | The difference in P1NP between treatment arms after 10 weeks
  The interaction between treatment and time on serum P1NP
Serum P1NP | The difference in P1NP between treatment arms after 12 weeks
  The interaction between treatment and time on serum P1NP
Serum P1NP | The difference in P1NP between treatment arms after 14 weeks
  The interaction between treatment and time on serum P1NP
Serum P1NP | The difference in P1NP between treatment arms after 16 weeks
  The interaction between treatment and time on serum P1NP

SECONDARY OUTCOMES:
Serum CTX | The difference in CTX between treatment arms after 2 weeks
  The interaction between treatment and time on serum CTX
Serum CTX | The difference in CTX between treatment arms after 4 weeks
  The interaction between treatment and time on serum CTX
Serum CTX | The difference in CTX between treatment arms after 6 weeks
  The interaction between treatment and time on serum CTX
Serum CTX | The difference in CTX between treatment arms after 8 weeks
  The interaction between treatment and time on serum CTX
Serum CTX | The difference in CTX between treatment arms after 10 weeks
  The interaction between treatment and time on serum CTX
Serum CTX | The difference in CTX between treatment arms after 12 weeks
  The interaction between treatment and time on serum CTX
Serum CTX | The difference in CTX treatment arms after 14 weeks
  The interaction between treatment and time on serum CTX
Serum CTX | The difference in CTX between treatment arms after 16 weeks
  The interaction between treatment and time on serum CTX

OTHER OUTCOMES:
Fasting glucose | The difference between treatment arms in terms of change in fasting glucose after 16 weeks
  Change in fasting glucose
Fasting insulin | The difference between treatment arms in terms of change in fasting insulin after 16 weeks
  Change in fasting insulin
Fasting insulin insulin resistance (HOMA-IR), and post-OGTT outcomes from to baseline until 16 weeks of treatment. | The difference between treatment arms in terms of change in HOMA-IR after 16 weeks
  Change in fasting insulin
Glucose levels after an oral glucose tolerance test (OGTT) | The difference between treatment arms in terms of change in post-OGTT glucose values after 16 weeks
  Change in glucose levels 2 hours after an oral glucose tolerance test (OGTT)
Change in liver steatosis | The difference between treatment arms in terms of change in CAP scores after 16 weeks
  Controlled Attenuation Parameter (CAP) scores, assessed with a Fibroscan

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Bisschop, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No